CLINICAL TRIAL: NCT04824924
Title: A Phase 2 Study of Venetoclax in Combination With Low-dose HHT, G-CSF, and AZA as First-line Treatment for Newly Diagnosed Elderly AML Patients Unfit for Intensive Chemotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Yang SHEN, Clinical professor, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YangSHEN
Record Dates: First submitted 2021-03-28; First posted 2021-04-01 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: AML; venetoclax; combination therapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HVAG regimen (Experimental)
  Interventions: Drug: The combination of HHT, venetoclax, AZA, G-CSF

INTERVENTIONS:
Drug: The combination of HHT, venetoclax, AZA, G-CSF — HVAG regimen in a 28-day cycle HHT: d1-d7 1mg/m2; VEN: d1 100mg, d2 200mg, d3-d28 400mg; AZA: d1-d7 75mg/m2; G-CSF: d1-d7 300mg

SUMMARY:
Acute myeloid leukemia (AML) is a group of heterogeneous malignancies derived from hematopoietic precursors. Patients older than 65 years can hardly benefit from standard intensive chemotherapy while having a poor toxicity tolerance, leading to a dismal prognosis. Currently, there is no satisfactory treatment modality for this high-risk patient population, which is an unmet clinical need.

Venetoclax (ABT-199/GDC-0199, VEN) is a highly selective, oral B-cell lymphoma 2 (BCL-2) inhibitor that has shown activity in BCL-2- dependent leukemia and lymphoma cell lines, and has recently exerted encouraging therapeutic effect with manageable toxicity profile in the field of treatment of AML. Promising results have emerged in the combination of venetoclax and hypomethylating agents (HMA), decitabine or azacitidin (AZA), producing complete remission (CR) plus CR with incomplete hematologic recovery (CRi) rates of 74% and 66.7%, respectively, in previously untreated elderly AML patients.

Homoharringtonine (HHT) is an alkaloid and has been used in Chinese patients with acute and chronic myeloid leukemia for more than 30 years. The add of HHT to the combination of cytarabin and aclarubicin or daunorubicin has been proved to improve CR rate and prognosis of AML patients. Moreover, HHT combined with low-dose cytarabine and granulocyte colony-stimulating factor (G-CSF) has achieved durable efficacy in AML patients, either in the first-line or salvage setting. Interestingly, HHT has potent synergistic effects with VEN through reducing the expression of BCL-XL and MCL-1 in BCL-2 related pathways as previouly reported.

This study aims at investigating the combination of HHT, VEN, AZA and G-CSF (HVAG) in the treatment of newly diagnosed elderly AML patients who are ineligible for intensive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have confirmation of Acute Myeloid Leukemia (AML) by World Health Organization (WHO) criteria, previously untreated and unfit for intensive chemotherapy
* Participant must be >= 60 years of age.
* Participant must have a projected life expectancy of at least 12 weeks.
* Participant must have adequate renal function as demonstrated by a creatinine >= 30 mL/min;determined via urine collection for 24-hour creatinine clearance or by the Cockcroft Gault formula
* Participant must have adequate liver function as demonstrated by:

  1. aspartate aminotransferase (AST) <= 3.0 x ULN*
  2. alanine aminotransferase (ALT) <= 3.0 x ULN*
  3. bilirubin <= 1.5 x ULN* * Unless considered to be due to leukemic organ involvement i. Subjects who are < 75 years of age may have a bilirubin of <= 3.0 x ULN

Exclusion Criteria:

* Participant has history of myeloproliferative neoplasm (MPN) including myelofibrosis, essential thrombocythemia, polycythemia vera, chronic myeloid leukemia (CML) with or without BCR-ABL1 translocation and AML with BCR-ABL1 translocation
* Participant has acute promyelocytic leukemia
* Participant has known active central nervous system (CNS) involvement with AML
* Participant is known to be positive for hepatitis B or C infection
* Participant has received anticancer therapies including chemotherapy, radiotherapy or other investigational therapy, including targeted small molecule agents within 5 half-lives prior to first dose of study drug
* Participant has received biologic agents (e.g. monoclonal antibodies) for anti-neoplastic intent within 30 days prior to first dose of study drug
* Participant has received the following within 7 days prior to the first dose of the study drug:

  1. Steroid therapy for anti-neoplastic intent;
  2. Strong and Moderate CYP3A inhibitors (see Appendix A for examples)
  3. Strong and Moderate CYP3A inducers (see Appendix A for examples)
* Participant exhibits evidence of other clinically significant uncontrolled systemic infection requiring therapy
* Participant has a serious cardiovascular, pulmonary or renal disability
* Participant has a history of other malignancies within 2 years prior to study entry, with the exception of:

  1. Adequately treated in situ carcinoma of the cervix uteri or carcinoma in situ of breast;
  2. Basal cell carcinoma of the skin or localized squamous cell carcinoma of the skin;
  3. Previous malignancy confined and surgically resected (or treated with other modalities) with curative intent; requires discussion with TA MD.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Rate of complete remission (CR) | Up to 36 months
  including Complete Remission with incomplete Platelet recovery (CRp) and Complete Remission with incomplete hematologic recovery (CRi)

SECONDARY OUTCOMES:
Event-free survival (EFS) | Up to 36months
  EFS is defined as the time from the date of randomization until the date of documented relapse or discontinuation of the treatment, or initiation of other anti-leukemic treatment or death from any cause, whichever occurs first
Relapse-free survival | 36 months
  Relapse-free survival (RFS) will be measured from time of CR to either leukemia relapse or death, whichever comes first. Leukemia relapse will be defined as bone marrow (BM) blasts 5% or higher (not attributable to regenerating BM), any circulating blasts (not attributable to regenerating BM or growth factors), or any extra-medullary blast foci as per Revised International Working Group (R-IWG) criteria.
Overall survival(OS) | Up to 36 months
Safety and tolerability assessed by incidence and severity of adverse events | 36 months
  All grade ≥ 3 toxicities according to CTCAE (Common Terminology Criteria for Adverse Events) version 5 will be tabulated

IPD SHARING:
Plan to Share IPD: No